CLINICAL TRIAL: NCT05518357
Title: An Exploratory Clinical Study on the Safety and Efficacy of LILRB4 STAR-T Cells in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
Brief Title: LILRB4 STAR-T Cells in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS104-001
Record Dates: First submitted 2022-07-04; First posted 2022-08-26 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LILRB4 STAR-T (Experimental): LILRB4 STAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of STAR-T cells, subjects receive fludarabine at dose 25-30mg/m2/day and cyclophosphamide treatment at dose 250-300mg/m2 for 3 days and take a rest for 2 days before infusion. STAR-T cells will be intravenously infused with a escalated dose of 1E6#3E6#1E7 cells/kg
  Interventions: Biological: LILRB4 STAR-T

INTERVENTIONS:
Biological: LILRB4 STAR-T — Subjects with relapsed/refractory acute myeloid leukemia will be enrolled in the study, and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of STAR-T cells. STAR-T cells will be intravenously infused with a escalated dose of 1E6#3E6#1E7 cells/kg。

SUMMARY:
This is a single-center, single-arm, open-label phase I clinical study to determine the safety and efficacy of LILRB4 STAR-T cells in relapsed/refractory acute myeloid leukemia subjects.

DETAILED DESCRIPTION:
This study will recruit LILRB4 positive AML subjects,and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of LILRB4 STAR-T cells. LILRB4 STAR-T cells will be intravenously infused with a escalated dose of 1E6、3E6、1E7 cells/kg.The purpose of current study is to evaluate the clinical safety and tolerability of LILRB4 STAR-T cells therapy in patients with refractory and relapsed AML.Safety and efficacy of LILRB4 STAR-T cells therapy will be monitored.The primary endpoint of the study is to observe DLT, AE, SAE, CRS and ICANS. Secondary objectives are to observe the efficacy of LILRB4 STAR-T cells, including RFS, EFS and OS, and PK.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2-70 years, gender is not limited;
2. Subjects diagnosed with AML according to WHO 2016 criteria and according to the "Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory Acute Myeloid Leukemia (2021 Edition)" should meet any of the following relapsed and refractory (R/R) AML patients:

   1. Patients who have failed two cycles of standard chemotherapy;
   2. Relapse within 12 months after consolidation and intensification therapy after complete remission (CR);
   3. Relapse after 12 months but failed to respond to conventional treatment
   4. two or more recurrences;
   5. persistent extramedullary leukemia；
3. ECOG physical status level is 0 to 2;
4. Bone marrow sample must be LILRB4 positive(Flow Cytometry)
5. Major organs must meet the following criteria:

   1. Liver function: Total bilirubin≤1.5 times the upper limit of normal,ALT and AST≤3 times the upper limit of normal,
   2. Renal function:Creatinine≤1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥60ml/min,
   3. Cardiac function:LVEF≥50%，
   4. Lung function:Defined as ≤grade 1 dyspnea and blood oxygen saturation >92%;
6. Female subjects of reproductive age or male subjects whose partners are women of reproductive age agree to use an effective method of contraception throughout the trial and for 12 months after cell infusion;
7. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Received CAR-T therapy or other gene-modified cell therapy in the past or participated in other clinical investigators within 1 month before screening;
2. Any of the following cardiovascular and cerebrovascular diseases occurred within 6 months before screening:

   1. congestive heart failure(NYHA stage III),myocardial infarction,unstable angina pectoris,congenital long QT syndrom,Anterior left block,coronary angioplasty,stent implantation,Coronary/peripheral artery bypass grafting,CVA,Transient ischemic attack or pulmonary embolism,Asymptomatic right bundle branch block was allowed;
   2. Serious arrhythmias requiring treatment (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, etc.);
   3. uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), a history of hypertensive crisis or hypertensive encephalopathy;
3. The subject is positive for hepatitis B surface antigen or HBV DNA is higher than the detection limit of analysis method;Positive hepatitis C antibody or HCV RNA is higher than the detection limit of the analytical method;The subjects were positive for syphilis antibody;
4. The subject with known systemic lupus erythematosus, active or uncontrolled autoimmune disease (such as Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.), primary or secondary immunodeficiency (such as HIV infection or serious infectious disease, etc.);
5. Previous or concurrent other incurable malignancies with unstable control,Affect the long-term survival of subjects, except for cured cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer or other local prostate cancer after radical treatment, ductal carcinoma in situ after radical resection and at least 5 Years without recurrence of malignant tumor;
6. Subjects with current or previous history of central nervous system disease, such as seizures, stroke, severe brain injury, aphasia, paralysis, dementia, Parkinson's disease, mental illness, etc. or central nervous system leukemia (CNSL);
7. Subjects with a history of solid organ transplantation or hematopoietic stem cell transplantation (HSCT) within 6 months prior to screening;
8. Subjects with aGVHD and cGVHD at screening;
9. Subjects who have had any of the following drugs or treatments within the specified time period prior to apheresis:

   1. Administered any immunosuppressant within 2 weeks prior to apheresis;
   2. Received any chemotherapy within 2 weeks or 3 half-lives, whichever is shorter, prior to apheresis;
   3. Received any macromolecule or small molecule targeted therapy such as monoclonal antibody, antibody-drug conjugate (ADC), double antibody, etc. within 4 weeks before apheresis or within 3 half-lives (whichever is shorter);
10. Those with mental illness or history of drug abuse;
11. Pregnant or breastfeeding subjects;
12. The investigator believes that there are other factors that are not suitable for inclusion or that affect subjects participating in or completing the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability | 12 months
  Subjects are observed for dose-limiting toxicity(DLT) after LILRB4 STAR-T cells infusion, with the recording of adverse events(AE) and serious adverse events(SAE), with a focus on cytokine release syndrome(CRS) and immune cell-associated neurotoxicity(ICANS).All of the AE ratings were assessed according to the CTCAE.

SECONDARY OUTCOMES:
Antitumor efficacy | 12 months
  After infusion of LILRB4 STAR-T cells, the subjects underwent bone marrow puncture every month to evaluate the tumor load in the bone marrow. The efficacy evaluation included complete morphological remission, complete remission with incomplete recovery of blood cytology, and partial remission.

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD/PHD, Principal Investigator — HeiBei YanDa Ludaopei hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China

IPD SHARING:
Plan to Share IPD: No